CLINICAL TRIAL: NCT05160415
Title: A Phase 1b, Open-label Study of the Safety and Pharmacokinetics of EDG-5506 in Adults With Becker Muscular Dystrophy
Brief Title: A Study of EDG-5506 in Adult Males With Becker Muscular Dystrophy
Acronym: ARCH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDG-5506-002
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Becker Muscular Dystrophy
Keywords: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Drug: Sevasemten
  Interventions: Drug: Sevasemten

INTERVENTIONS:
Drug: Sevasemten — Daily oral dose of 10 mg daily until Visit 8 (Day 57), followed by 15 mg daily until Visit 13 (Month 6), followed by 20 mg until Visit 21 (Month 15), followed by 10 mg daily to Visit 27 (Month 24).
  Other Names: EDG-5506

SUMMARY:
The ARCH study was an open-label, single-center, Phase 1b study of sevasemtem (EDG-5506) to assess the safety and pharmacokinetics (PK) of sevasemten in adults with Becker muscular dystrophy (BMD).

Sevasemten is an investigational product intended to protect and improve function of dystrophic muscle fibers.

DETAILED DESCRIPTION:
This open-label study evaluated the safety, tolerability, and pharmacokinetics (PK) of sevasemten in participants with BMD who completed the first-in-human study, EDG-5506-001, as well as additional (treatment-naïve) participants from outside the EDG-5506-001 study to meet the target sample size.

All participants received sevasemten. This study had a 24 month treatment period, followed by an optional 4 week follow-up period. On-site visits occurred approximately monthly for the first 12 months, followed by every 3 months to assess safety and measures of function.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have completed Study EDG-5506-001.
2. Participants who were not from Study EDG-5506-001 must meet the following:

   1. Male sex at birth and aged 18 to 55 years inclusive at time of consent.
   2. Documented dystrophin mutation with phenotype consistent with BMD.
   3. Ambulatory at Screening (defined as ability to complete 100 meter [m] timed test, with or without assistance).
   4. Body weight ≥ 50 kg at the Screening visit.
   5. Body mass index (BMI) between 20 and 34 kg/m2 inclusive.
3. Female sexual partners of male participants must use highly effective contraception (<1% failure rate per year) through 6 months after last dose.
4. Capable of giving signed informed consent.

Exclusion Criteria:

1. Any clinically significant changes during or following the completion of Study EDG 5506-001 that would affect the potential safety of the participant to receive EDG 5506.
2. Cardiac echocardiogram ejection fraction <45% or New York Heart Association (NYHA) Class III or Class IV.
3. Baseline 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
4. Forced vital capacity (FVC) predicted <65% or using daytime (mechanical or noninvasive) ventilatory support.
5. Moderate or severe renal or hepatic impairment (eGFR <60 mL/min/1.73 m2).
6. Positive test for hepatitis C antibody (unless negative HCV PCR), hepatitis B surface antigen, or human immunodeficiency virus (HIV) antibody at screening.
7. History of substance abuse or dependency.
8. Receipt of oral corticosteroids for >5 days in the previous 6 months at a dose of >5 mg equivalent per day. Lower oral doses or inhaled/intranasal steroids are permitted.
9. Receiving moderate or strong cytochrome P450 CYP3A4 inhibitors or inducers.
10. Participation in any other investigational drug study or use of use of an investigational drug within 30 days or 5 half-lives (whichever is longer) of dosing in the present study.
11. Participants who are unlikely to comply with the study protocol or, in the opinion of the Investigator, would not be a suitable candidate for participation in the study.
12. Medical history or other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory result or abnormality that may increase the risk of study participation or, in the Investigator's judgment, make the participant inappropriate for the study. Includes venous access that would be too difficult to facilitate repeated blood sampling.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rare Disease Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.edgewisetx.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 12
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Height [Mean (Standard Deviation); unit: cm] | 175.37 (6.747)
Weight [Mean (Standard Deviation); unit: kg] | 77.77 (10.563)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Treated With Sevasemten Experiencing AEs
Description: An AE is any untoward medical occurrence in a patient administered a medicinal product. The AE does not necessarily have to have a causal relationship with the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  The numerator of the percentage is the number of participants experiencing at least one AE after first dose of study drug up to 25 months.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants | 100

2. Primary Outcome: Frequency of AEs in Those Treated With Sevasemten
Description: An AE is any untoward medical occurrence in a patient administered a medicinal product. The AE does not necessarily have to have a causal relationship with the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  The endpoint is the cumulative total number of AEs occurring after first dose of study drug up to 25 months among participants who received at least one dose of study drug.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: Count of Events
Arm/Group | Treatment
Number analyzed (Participants) | 12
Count of Events | 95

3. Primary Outcome: Number of Participants Treated With Sevasemten With AEs by Maximum Severity
Description: An AE is any untoward medical occurrence in a patient administered a medicinal product. The AE does not necessarily have to have a causal relationship with the study drug. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  The severity of an AE is graded, according to the study protocol definitions of AE severity/intensity, as "mild", "moderate" or "severe". Participants who reported multiple AEs are counted only once at the highest severity reported.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants
  Mild | 10
  Moderate | 2
  Severe | 0

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Abnormal Clinical Chemistry Test Results
Description: Treatment-emergent defined as any event that occurs after the start of study drug or was present at baseline and worsened after taking study drug.
  The numerator of the percentage is the number of participants experiencing at least one treatment-emergent abnormal clinical chemistry test result after first dose of study drug up to 25 months.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants | 0

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Abnormal Hematology Test Results
Description: Treatment-emergent defined as any event that occurs after the start of study drug or was present at baseline and worsened after taking study drug.
  The numerator of the percentage is the number of participants experiencing at least one treatment-emergent abnormal hematology test result after first dose of study drug up to 25 months.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants | 0

6. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Abnormal Coagulation Test Results
Description: Treatment-emergent defined as any event that occurs after the start of study drug or was present at baseline and worsened after taking study drug.
  The numerator of the percentage is the number of participants experiencing at least one treatment-emergent abnormal coagulation test result after first dose of study drug up to 25 months.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants | 0

7. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Abnormal Urinalysis Test Results
Description: Treatment-emergent defined as any event that occurs after the start of study drug or was present at baseline and worsened after taking study drug.
  The numerator of the percentage is the number of participants experiencing at least one treatment-emergent abnormal urinalysis test result after first dose of study drug up to 25 months.
Time Frame: From first dose of study drug to 25 months
Population: Participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of participants | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry
Description: Refer to Protocol for list of clinical chemistry tests that were performed. Clinically significant changes in clinical chemistry are defined as adverse events related to clinical chemistry tests or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology
Description: Refer to Protocol for list of hematology tests that were performed. Clinically significant changes in hematology are defined as adverse events related to hematology tests or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Coagulation
Description: Refer to Protocol for list of coagulation tests that were performed. Clinically significant changes in coagulation are defined as adverse events related to coagulation tests or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Refer to Protocol for list of urinalysis tests that were performed. Clinically significant changes in urinalysis are defined as adverse events related to urinalysis tests or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Supine systolic and diastolic blood pressure, pulse rate, respiratory rate, and temperature were measured. Clinically significant changes in vital signs are defined as adverse events related to vital signs or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Physical and Neurological Examinations
Description: A physical examination included head, ears, eyes, nose, mouth, skin, heart and lung, lymph nodes, and gastrointestinal and musculoskeletal systems. A neurological examination was also conducted to include upper and lower limb tone, power, reflexes, and examination of cranial nerves II-XII (excluding ophthalmoscopy). Clinically significant changes in physical and neurological examinations are defined as adverse events related to physical and neurological examinations or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in ECG PR Interval
Description: Triplicate 12-lead electrocardiogram (ECG) parameters were obtained using an ECG machine that automatically measured PR interval. Clinically significant changes in ECG PR interval are defined as adverse events related to ECG PR interval or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Changes in ECG QRS Interval
Description: Triplicate 12-lead electrocardiogram (ECG) parameters were obtained using an ECG machine that automatically measured QRS interval. Clinically significant changes in ECG QRS interval are defined as adverse events related to ECG QRS interval or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Changes in ECG QT Interval
Description: Triplicate 12-lead electrocardiogram (ECG) parameters were obtained using an ECG machine that automatically measured QT interval. Clinically significant changes in ECG QT interval are defined as adverse events related to ECG QT interval or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Changes in ECG QTc Interval
Description: Triplicate 12-lead electrocardiogram (ECG) parameters were obtained using an ECG machine that automatically measured QT corrected (QTc) Interval. QT corrected by Bazett's formula (QTcB) and QT corrected by Fridericia's formula (QTcF) were both recorded. Clinically significant changes in ECG QTc interval are defined as adverse events related to ECG QTc interval or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Changes in Forced Vital Capacity (FVC)
Description: Assessed by spirometry. Clinically significant changes in FVC are defined as adverse events related to FVC or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Changes in Forced Expiratory Volume in 1 Second (FEV1)
Description: Assessed by spirometry. Clinically significant changes in FEV1 are defined as adverse events related to FEV1 or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Changes in Cardiac Function as Assessed by Echocardiogram
Description: Echocardiographic examinations were performed by a qualified individual (sonographer) at the site to evaluate left-ventricular systolic and diastolic function, geometry, and mass, as well as left-atrial and right-ventricular function and geometry via two-dimensional, doppler, and/or speckle-tracking imaging techniques. Valvular competence, including presence or absence of regurgitation, was evaluated and quantified, while overall cardiac health was qualitatively evaluated (e.g., presence/absence of pericardiac effusion).
  Clinically significant changes in cardiac function are defined as adverse events related to cardiac function as assessed by echocardiogram or investigator identified results reported from first dose of study drug up to 24 months. Only clinically significant changes were counted.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Changes in Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a questionnaire used for suicide assessment. The assessment includes "yes" or "no" responses for 6 questions. Questions 1-5 are related to suicidal ideation, including: 1=Wish to be Dead, 2=Non-specific Active Suicidal Thoughts, 3=Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act, 4=Active Suicidal Ideation with Some Intent to Act, without Specific Plan, 5=Active Suicidal Ideation with Specific Plan and Intent. Question 6 is related to suicidal behavior and asks about actual attempts. Numeric ratings were provided for severity of ideation (if present), from 1 to 5, with 5 being the most severe. For this study, clinically significant changes in C-SSRS are defined as responses of "yes" to suicidal ideation or suicidal behavior item as measured by C-SSRS or investigator identified results reported from first dose of study drug to 24 months.
Time Frame: From first dose of study drug to 24 months
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 12
Participants | 0

22. Secondary Outcome: Plasma Sevasemten (EDG-5506) Concentrations at Sample Timepoints
Description: Values below the limit of quantitation (BLQ) of 0.500 ng/mL were treated as 0 before the first quantifiable concentration and as missing elsewhere.
  Single PK concentration was collected at each visit, except for Day 1. For treatment-naive participants, Day 1 was a serial collection at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 24 hours post-dose. The last timepoint was on Day 2. The dose on Day 2 was administered only after the 24 hour timepoint. For treatment experienced participants, Day 1 was pre-dose only.
  Days 29 and 57 have window of +/- 3 days; Months 3-24 have window of +/- 5 days.
Time Frame: Pre-dose; 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 24 hours post-dose; 29 and 57 days post-dose; 3, 4, 6, 7, 8, 10, 12, 15, 18, 21, and 24 months post-dose.
Population: Participants who received at least one dose of study drug and have a sufficient PK profile to derive at least one PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment
Number analyzed (Participants) | 12
ng/mL
  Pre-dose: number analyzed (Participants) | 10
  Pre-dose | 0 (0)
  0.25 hours: number analyzed (Participants) | 6
  0.25 hours | 3.671 (4.1099)
  0.5 hours: number analyzed (Participants) | 7
  0.5 hours | 23.19 (30.408)
  1 hour: number analyzed (Participants) | 7
  1 hour | 21.68 (15.091)
  1.5 hours: number analyzed (Participants) | 7
  1.5 hours | 22.57 (10.959)
  2 hours: number analyzed (Participants) | 7
  2 hours | 21.60 (18.013)
  3 hours: number analyzed (Participants) | 7
  3 hours | 12.63 (6.5033)
  4 hours: number analyzed (Participants) | 7
  4 hours | 8.899 (2.3685)
  6 hours: number analyzed (Participants) | 7
  6 hours | 6.536 (2.5716)
  24 hours: number analyzed (Participants) | 7
  24 hours | 4.000 (1.5452)
  29 days | 53.27 (20.607)
  57 days | 60.57 (26.389)
  3 months | 93.63 (38.939)
  4 months: number analyzed (Participants) | 11
  4 months | 92.34 (34.940)
  6 months | 105.3 (40.764)
  7 months | 137.4 (52.673)
  8 months | 137.7 (55.542)
  10 months | 149.3 (69.139)
  12 months | 141.7 (60.399)
  15 months: number analyzed (Participants) | 10
  15 months | 175.2 (58.905)
  18 months: number analyzed (Participants) | 9
  18 months | 78.20 (34.885)
  21 months: number analyzed (Participants) | 10
  21 months | 69.33 (26.315)
  24 months: number analyzed (Participants) | 10
  24 months | 55.38 (29.536)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 25 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=12)
COVID-19 (Infections and infestations) | 5
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 3
Arthropod sting (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Gait inability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Testicle adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT05160415/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT05160415/SAP_001.pdf